CLINICAL TRIAL: NCT02012400
Title: Effects of Regular Exercise on Physical Fitness, Asthma Control and Quality of Life of Adult Asthmatics
Brief Title: Effects of Regular Exercise on Adult Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: GlaxoSmithKline (Industry); Foundation of the Finnish Anti-Tuberculosis Association (Unknown); Research Foundation of the Pulmonary Diseases (Unknown); Jalmari and Rauha Ahokas Foundation (Unknown); Vaino and Laina Kivi Foundation (Unknown); Ida Montini Foundation (Other); Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mjaakkola-001
Record Dates: First submitted 2013-05-30; First posted 2013-12-16 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Asthma; Exercise; Asthma control; Physical fitness; Quality of life
MeSH Terms: conditions — Asthma; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Exercise
- Control group (No Intervention)

INTERVENTIONS:
Other: Exercise — The exercise group is given a 24-week individualized training program, including aerobic exercise, muscular training, relaxation exercises and stretching. Patients are asked to observe their asthma control daily and to mark in their diary asthma symptoms and activity limitations as well as duration, intensity and form of exercising on daily basis. They are also asked to perform PEF-measurements twice a day for one-week period every 4 weeks. The control group receives ordinary instructions.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to assess the effects of regular exercise on physical fitness, asthma control, and quality of life among adult asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of asthma made by physician, or reimbursement for asthma medication from the National Social Insurance Institution of Finland (code 203), or patient fulfills the diagnostic criteria for asthma as outlined in the Finnish Guidelines for Asthma Management (Käypä hoito -suositus 2006 and 2012)

Exclusion Criteria:

* FEV1 < 60 % of predicted in spirometry
* PEF variability > 30 % at least 2 times during a 1-week monitoring period
* use of bronchodilating medication at least 4 times daily
* permanent, daily steroid tablet treatment
* patients who exercise regularly already at baseline at least 3 times a week at least 30 min at a time
* serious coronary heart disease
* severe hypotension
* severe heart failure
* severe musculoskeletal disorder
* dementia
* physician-diagnosed chronic obstructive lung disease

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Asthma control | 6-month period
  Asthma control based on symptom score and PEF-values

SECONDARY OUTCOMES:
Physical fitness | Baseline and 6 months
  Physical fitness measured with spiroergometry

OTHER OUTCOMES:
Lung function | Baseline and 6 months
  Lung function measured with spirometry
Quality of Life | Baseline and 6 months
  Quality of life assessed using St. Georges Respiratory Questionnaire
Step test | Baseline and 6 months
  Indirect maximal oxygen consumption test using with 6 min step-walk-test
Muscle strength and flexibility | Baseline and 6 months
  Muscle strength and flexibility tests

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Environmental and Respiratory Health Research, University of Oulu, Oulu, Finland